CLINICAL TRIAL: NCT02822807
Title: Q Fever and Auto-immunity
Acronym: Q Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-31; 2013-A00963-42 (Other: ANSM)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2022-10

CONDITIONS: Q Fever; Auto-Immunity
MeSH Terms: conditions — Q Fever | interventions — Blood Specimen Collection

ARMS (4):
- Q fever without valvular disease (Other): Q fever without valvular disease
  Interventions: Biological: Blood sampling
- Q fever with valvular disease (Other): Q fever with valvular disease
  Interventions: Biological: Blood sampling
- Q fever infective endocarditis (Other): Q fever infective endocarditis
  Interventions: Biological: Blood sampling
- Other Coxiella burnetii infections (including pregnant women) (Other): Other Coxiella burnetii infections (including pregnant women)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling

SUMMARY:
The IHU Mediterranean infection is national reference centre for Q fever. Coxiella burnetii is the bacteria responsible of this infection. The bacterium Coxiella burnetii infection is associated with secretion by the body both many antibodies against the bacteria but also against certain cells of the body (autoantibodies). These autoantibodies may have no effect or be associated with specific symptoms. Anti-Phospholipid antibodies are especially prevalent in the Q fever. Apart from this infection, they are associated with thrombocytopenia, obstetric complications, thrombosis and heart valve damage. These conditions have also been described as complications during Q fever. In a retrospective preliminary work on Q fever, we have shown that the presence of high levels of IgG anti-cardiolipin was associated with the presence of valvular and the evolution to endocarditis. Such associations have a therapeutic involvement and must therefore be confirmed. Indeed, if these associations were confirmed, a trans-esophageal ultrasound could be systematically proposed to patients with valvular disease of trans-thoracique ultrasound but IgG anticardiolipin high levels. Other special attention could be given to patients with high autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a current or former Q fever diagnosis
* Patient > or = 18 years old.
* Patient who does not declined to have his medical records reviewed for research.
* Patient with health insurance.

Exclusion Criteria:

* Minor patient (<18 years )
* Adult patient under guardianship .
* Patient deprived of liberty or judgment.
* Patient refusing to sign the informed consent form .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of a complication, linked to the rate of autoantibodies. | 2 years
  The required complications are the followings:
  * endocarditis
  * thrombosis
  * thrombocytopenia
  * obstetrical complications:
    * Spontaneous miscarriage defined as a spontaneous expulsion of the embryo before 20 weeks gestation .
    * Spontaneous abortion
    * Fetal intrauterine death
    * Oligoamnios
    * Intrauterine growth retardation
    * Fetal malformations .

SECONDARY OUTCOMES:
Rate of anti- cardiolipin antibodies | 1 day
Rate of anti- phagosome autoantibodies | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Didier RAOULT, PR, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France